CLINICAL TRIAL: NCT02443363
Title: Estimated Glomerular Filtration Rate After Kidney Transplantation - the Formula Modification of Diet in Renal Disease (MDRD), Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) or Cockroft-Gault?
Brief Title: Estimated Glomerular Filtration Rate After Kidney Transplantation - the Formula MDRD, CKD-EPI or Cockroft-Gault?
Acronym: eGFR
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Czyżewski, Łukasz Czyżewski, Medical University of Warsaw
Other Study IDs: GFR/KTx/2015/04
Record Dates: First submitted 2015-05-10; First posted 2015-05-13 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Renal Function Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients After Kidney Transplantation: A total of 300 consecutive patients admitted to routine visit in Transplant Centre with functioning graft longer than 3 months to 10 years
  Interventions: Other: Estimating of formula MDRD, CKD-EPI, Cockroft-Gault,; Device: Tanita BC 418- Bioelectrical impedance analysis

INTERVENTIONS:
Other: Estimating of formula MDRD, CKD-EPI, Cockroft-Gault,
Device: Tanita BC 418- Bioelectrical impedance analysis — The device measured the size of total body water (TBW), fat mass (FM%), visceral fat%, fat free mass (FFM), and basal metabolic rate (BMR) (kcal).

SUMMARY:
The study included 300 patients who are post-kidney transplantation (> 3 months and <10 years). An analysis of body composition using bioelectrical impedance, calculated BMI and serum creatinine was determined. Glomerular filtration rate (GFR) was calculated using the formula CKD-EPI, Modification of Diet in Renal Disease (MDRD) and Cockroft-Gault.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* functioning graft longer than 3 months to 10 years
* no clinical cardiovascular disease during the 6 months preceding entry
* stable graft function- glomerular filtration rate > 30 ml/min/1.73 m2, creatinine concentration <2.5 mg/dl

Exclusion Criteria:

* not meet the above criteria
* episode of illness (for example: infection)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 consecutive patients after kidney transplantation admitted to routine visit in Transplant Centre
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Differences in estimating GFR using formula MDRD, CKD-EPI and Cockroft-Gault in short and long-term postoperative period. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Mazovian, Poland